CLINICAL TRIAL: NCT02882555
Title: Effect of Muscular Exercise on Cough Reflex
Acronym: REFLEXE TOUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-A00390-57
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Exercise; Capsaicin; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children (Experimental): 12 concentrations of caspaicin are administered: - 0.6, 1.2, 2.4, 4.8, 9.8, 19.5, 39, 78.1, 156.2, 312.5, 625, 1250 μmol/l. Capsaicin concentration eliciting at least 2 coughs (C2) or 5 coughs (C5) is determined.
  At least 1-hour-interval from capsaicin dose titration (in order to minimize tachyphylaxy)
  Administration of 4 inhalations at 1-min-interval: 2 C5 and 2 controls (normal saline) in random order at baseline
  At least 1-hour-interval (in order to minimize tachyphylaxy)
  Administration of 4 inhalations at 1-min-interval: 2 C5 and 2 controls in random order during exercise, when heart rate is maximum
  Interventions: Behavioral: Exercise; Drug: Capsaicin; Drug: Normal saline
- Adults (Active Comparator): As reference for more precise assessment of effects of development.
  12 concentrations of caspaicin are administered: 0.49, 0.98, 1.95, 3.9, 7.8, 15.6, 31.3, 62.5, 125, 250, 500, 1000 μmol/l. Capsaicin concentration eliciting at least 2 coughs (C2) or 5 coughs (C5) is determined.
  At least 1-hour-interval from capsaicin dose titration (in order to minimize tachyphylaxy)
  Administration of 4 inhalations at 1-min-interval: 2 C5 and 2 controls (normal saline) in random order at baseline
  At least 1-hour-interval (in order to minimize tachyphylaxy)
  Administration of 4 inhalations at 1-min-interval: 2 C5 and 2 controls in random order during exercise, when heart rate is maximum
  Interventions: Behavioral: Exercise; Drug: Capsaicin; Drug: Normal saline

INTERVENTIONS:
Behavioral: Exercise — 6 min running on a motor-driven tredmill in a climate room (18-20°C, humidity <10 mg/l). Tredmill speed and slope are adjusted to increase heart rate to about 80 % of maximum value predicted for age (= 210 - age in years) during the first 2-3 min and pursued until the end of exercise (3-4 min). Heart rate is measured during the whole exercise.
Drug: Capsaicin — A compressed air-driven nebuliser is controlled by a dosimeter and a valve is used to deliver similar inspiratory flows for 400 msec in children and 1200 msec in adults.
Drug: Normal saline — A compressed air-driven nebuliser is controlled by a dosimeter and a valve is used to deliver similar inspiratory flows for 400 msec in children and 1200 msec in adults.

SUMMARY:
The hypothesis is that the cough reflex induced by capsaicin is inhibited during exercise. The purpose of this study is to determine if a short muscular exercise inhibits the cough reflex induced by capsaicin inhalation.

DETAILED DESCRIPTION:
Cough is an important reflex of defense of airways. It is also one of the more frequent symptoms during respiratory diseases. Chronic cough can be a disabling condition, apparently idiopathic or associated to pathology such as asthma, sinusitis with posterior discharge or gastroesophageal reflux.

Factors susceptible to provoke or increase cough are well known, but inhibiting factors are much less known. Muscular exercise is thought to influence respiratory reflexes in a considerable and complicated way. For example, a bronchodilation is observed in healthy or asthmatic individuals, but recovery period frequently triggers asthma attacks. Effects of exercise on cough reflex are much less known.

This study aims to determine the influence of muscular exercise on cough reflex in children and healthy adults.

Highlighting the inhibition of cough reflex by exercise can have a significant effect on chronic cough patient care. There is actually no symptomatic treatment really effective without side effects.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining of informed consent (or informed consent of parents or persons with parental authority)
* Affiliation to social security
* Negative answer to all 12 questions of medical questionnaire for child or to all 11 questions of medical questionnaire for adult
* Normal cardio-respiratory examination
* Normal electrocardiogram
* Without spirometry obstructive syndrome (FEV1 > 70% of predicted value and FEV1/FVC >70%)

Exclusion Criteria:

* Refusal or impossibility of obtaining informed consent of person or of persons with parental authority)

Ages: 7 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of cough efforts occurring within 15 sec of the C5 aerosol at baseline and during exercise | day 0
  Video-taped and identified from its sound by 2 observers

CONTACTS AND LOCATIONS:
Overall Officials: François MARCHAL, Pr, Principal Investigator — Explorations fonctionnelles pédiatriques, Hôpital d'enfants, CHRU de Nancy, France

IPD SHARING:
Plan to Share IPD: No